CLINICAL TRIAL: NCT02672462
Title: The Safety and Efficacy of a Renal Denervation System in Treating Patients With Hypertension: A Pilot Study
Brief Title: Renal Denervation for the Treatment of Hypertension: A Pilot Safety and Efficacy Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Golden Leaf MedTec Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GL-CT-20150301
Record Dates: First submitted 2016-02-01; First posted 2016-02-03 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

ARMS (1):
- Renal denervation (Experimental)
  Interventions: Device: Radio frequency renal denervation system (Golden Leaf GL-06E15A)

INTERVENTIONS:
Device: Radio frequency renal denervation system (Golden Leaf GL-06E15A)

SUMMARY:
A single center, self-controlled pilot study on safety and efficacy of renal denervation in treatment of hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Ages of 18 to 75, male or female;
* Main renal artery, with or without accessary renal arteries, with length

  * 20mm;
* Patients who have not taken any anti-hypertensive drugs or have been off drugs for at least 2 weeks, with mean SBP ≥150mmHg and

  * 180mmHg based on at least 3 office blood pressure measurements, or ASBP≥135mmHg and ≤170mmHg based on 24 hr blood pressure monitoring;
* Agrees to take part in the trial and signs the written, informed consent.

Exclusion Criteria:

* Renal artery abnormalities that are inappropriate for the procedure;
* Pregnant or plan to become pregnant;
* History of orthostatic hypotension;
* Type I diabetes;
* Estimated GFR<40mL/min/1.73m2;
* Only one kidney or prior kidney transplantation;
* Bleeding tendency or other coagulation related diseases;
* Acute or severe systemic infection;
* Prior renal artery interventional procedures or prior RDN treatment;
* History of stroke or TIA;
* Malignant tumor or end-stage illnesses;
* Secondary hypertension;
* Acute coronary events within 2 weeks;
* Other conditions that deem unsuitable for the procedure, in the opinions of investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
blood pressure | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gengshan Ma, MD, Principal Investigator — Cardiovascular division, Dept. of Internal Medicine, Zhongda Hospital
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China